CLINICAL TRIAL: NCT04389983
Title: Ketone Levels Achieved After Medium Chain Triglyceride (MCT) Oil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Angela Juby, PI, University of Alberta
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 00087958
Record Dates: First submitted 2020-05-07; First posted 2020-05-15 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Pharmacokinetics
Keywords: MCT oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy, under 65 years (Active Comparator): Four study days. Day 1 administered 0g MCT oil with baseline and hourly betahydroxybutyrate (BHB) measures (by fingerstick test) for 5 hours thereafter Day 2 administered 14g MCT oil with baseline and hourly betahydroxybutyrate (BHB) measures (by fingerstick test) for 5 hours thereafter Day 3 administered 28g MCT oil with baseline and hourly betahydroxybutyrate (BHB) measures (by fingerstick test) for 5 hours thereafter Day 4 administered 42g MCT oil with baseline and hourly betahydroxybutyrate (BHB) measures (by fingerstick test) for 5 hours thereafter (All MCT doses administered as a single dose at time 0)
  Interventions: Dietary Supplement: Medium Chain Triglyceride oil
- Healthy, over 65 years (Active Comparator): Four study days. Day 1 administered 0g MCT oil with baseline and hourly betahydroxybutyrate (BHB) measures (by fingerstick test) for 5 hours thereafter Day 2 administered 14g MCT oil with baseline and hourly betahydroxybutyrate (BHB) measures (by fingerstick test) for 5 hours thereafter Day 3 administered 28g MCT oil with baseline and hourly betahydroxybutyrate (BHB) measures (by fingerstick test) for 5 hours thereafter Day 4 administered 42g MCT oil with baseline and hourly betahydroxybutyrate (BHB) measures (by fingerstick test) for 5 hours thereafter.
  (All MCT doses administered as a single dose at time 0)
  Interventions: Dietary Supplement: Medium Chain Triglyceride oil
- Alzheimer's Disease subjects (Active Comparator): Four study days. Day 1 administered 0g MCT oil with baseline and hourly betahydroxybutyrate (BHB) measures (by fingerstick test) for 5 hours thereafter Day 2 administered 14g MCT oil with baseline and hourly betahydroxybutyrate (BHB) measures (by fingerstick test) for 5 hours thereafter Day 3 administered 28g MCT oil with baseline and hourly betahydroxybutyrate (BHB) measures (by fingerstick test) for 5 hours thereafter Day 4 administered 42g MCT oil with baseline and hourly betahydroxybutyrate (BHB) measures (by fingerstick test) for 5 hours thereafter.
  (All MCT doses administered as a single dose at time 0)
  Interventions: Dietary Supplement: Medium Chain Triglyceride oil

INTERVENTIONS:
Dietary Supplement: Medium Chain Triglyceride oil — Bulletproof Braine Octane MCT oil

SUMMARY:
Assessing Ketone levels achieved after varying doses of Medium Chain Triglyceride (MCT) oil

DETAILED DESCRIPTION:
Assessing Ketone levels achieved after varying doses of Medium Chain Triglyceride (MCT) oil in three study populations: <65 year healthy, 65 and older healthy, and Alzheimer's disease.

Each subject attends for 4 study days, receiving incrementally larger MCT doses at each visit for 0g, to 14g, to 28g to 42g.

ELIGIBILITY:
Inclusion Criteria:

* adult, healthy or with AD

Exclusion Criteria:

* unable to attend all study days
* coconut allergy
* Diabetes

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | 3 months
  Calculation of Cmax to varying doses in each subject and in different study arms.
Time to maximum plasma concentration (tmax) | 3 months
  Calculation of tmax to varying doses in each subject and in different study arms.
Area under the curve (AUC) | 3 months
  Calculation of AUC to varying doses in each subject and in different study arms.

SECONDARY OUTCOMES:
weight | 3months
  measured in kg
height | 3 months
  measured in cm
BMI | 3months
  Calculated BMI (ht/m2)
Body fat | 3 months
  % measured by bioimpedence scale

CONTACTS AND LOCATIONS:
Overall Officials: Angela Juby, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No